CLINICAL TRIAL: NCT05143567
Title: Comprehensive Assessment of the Hemostasis and Inflammation in Patients With Venous and Arterial Thrombotic Complications in Treatment of New Coronaviral Infection (COVID-19)
Brief Title: Hemostasis and Inflammation in COVID-19 Patients With Venous and Arterial Thrombotic Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Principal Investigator, Agapov Andrey Borisovich, Post-doctoral researcher, Ryazan State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11.10.2021
Record Dates: First submitted 2021-11-20; First posted 2021-12-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Venous Thromboembolism; covid19; Thrombosis
Keywords: venous thromboembolism; VTE; thrombotic events; coronavirus; COVID-19; hemostasis; platelet function
MeSH Terms: conditions — Venous Thromboembolism; COVID-19; Thrombosis; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Open-label cohort longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with COVID-19 without thrombotic complications (Experimental): Group I: 50 patients with confirmed coronavirus infection without thrombotic complications
  Interventions: Other: standard of care anticoagulation in absence of thrombotic complications
- patients with COVID-19 and VTE who received pharmacological prophylaxis of VTE (Experimental): Group II: 50 patients with confirmed coronavirus infection with thrombotic complications confirmed by ultrasonography with pharmacological prophylaxis of VTE
  Interventions: Other: standard of care anticoagulation in presence of thrombotic complications
- patients with COVID-19 and VTE who received pharmacomechanical prophylaxis of VTE (Experimental): Group III: 50 patients with confirmed coronavirus infection with ultrasound-confirmed thrombosis of the deep and saphenous veins of the lower extremities using pharmacomechanical prophylaxis of VTE.
  Interventions: Other: standard of care anticoagulation in combination with elastic compression

INTERVENTIONS:
Other: standard of care anticoagulation in absence of thrombotic complications — Subgroup IA - patients receive UFH (heparin, 7500 Units 2-3 times daily) for the prevention or treatment of VTE Subgroup IB - patients receive LMWH (enoxaparin) for the prevention or treatment of VTE Subgroup IC - patients receive oral anticoagulants (rivaroxaban 10mg QD) for the prevention or treatment of VTE
  Arms: patients with COVID-19 without thrombotic complications
Other: standard of care anticoagulation in presence of thrombotic complications — Subgroup IIA - patients receive UFH (heparin, 7500 Units 2-3 times daily) for the prevention or treatment of VTE Subgroup IIB - patients receive LMWH (enoxaparin, 0.4ml 2 times daily) for the prevention or treatment of VTE Subgroup IIC - patients receive oral anticoagulants (rivaroxaban 10mg QD) for the prevention or treatment of VTE
  Arms: patients with COVID-19 and VTE who received pharmacological prophylaxis of VTE
Other: standard of care anticoagulation in combination with elastic compression — Subgroup IIIA - patients receive UFH (heparin, 7500 Units 2-3 times daily) in combination with class II elastic compression (compression stockings above the level of the knee) for the prevention or treatment of VTE Subgroup IIIB - patients receive LMWH (enoxaparin, 0.4ml 2 times daily) in combination with class II elastic compression (compression stockings above the level of the knee) for the prevention or treatment of VTE Subgroup IIIC - patients receive oral anticoagulants (rivaroxaban 10mg QD) in combination with class II elastic compression (compression stockings above the level of the knee) for the prevention or treatment of VTE
  Arms: patients with COVID-19 and VTE who received pharmacomechanical prophylaxis of VTE

SUMMARY:
The study is aimed at assessing the role of the activity of high-risk markers of thrombotic events (MCP-1, MIP1α, IP-10, phosphatedylserine, calreticulin) on the development of thrombotic complications in patients with COVID -19.

DETAILED DESCRIPTION:
The study is aimed at assessing the role of the activity of high-risk markers for thrombotic events (monocytic chemoattractant protein 1 (MCP-1), macrophage inflammatory protein 1α (MIP1α), interferon-induced gamma protein-10 (IP-10), platelet apoptosis markers (phosphatedylserine, calreticulin) on the development of thrombotic complications in patients with COVID -19.

The study will include 150 patients of similar age, gender, and ethnicity, and they will be divided into three groups: Group I: 50 patients with confirmed coronavirus infection without thrombotic complications; Group II: 50 patients with confirmed coronavirus infection with thrombotic complications confirmed by ultrasonography without the use of pharmacomechanical prophylaxis of VTE; Group III: 50 patients with confirmed coronavirus infection with ultrasound-confirmed thrombosis of the deep and saphenous veins of the lower extremities using pharmacomechanical prophylaxis of VTE

ELIGIBILITY:
Inclusion Criteria:

* men or women over 18 years of age with a new coronavirus infection, confirmed by polymerase chain reaction (PCR) studies and chest CT.

Exclusion Criteria:

* men or women under 18 years of age; active cancer or a remission period of less than 5 years; decompensated somatic pathology; pregnancy or breastfeeding in women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
mortality | one year
  lethal outcomes
venous thrombosis or pulmonary embolism | one year
  a VTE event
arterial thrombosis | one year
  thrombosis of main arteries of the extremities or myocardial infarction or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Igor Suchkov, MD, PhD, Study Chair — Ryazan State Medical University
Locations (1):
- Ryazan State Medical University, Ryazan, Russia

IPD SHARING:
Plan to Share IPD: No